CLINICAL TRIAL: NCT03248115
Title: Bioavailability of Green Tea and Coffee Polyphenols in Healthy Participants
Brief Title: Bioavailability of Green Tea and Coffee Polyphenols
Acronym: POBAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MRC Human Nutrition Research (Other Government)
Responsible Party: Principal Investigator, Virginia Tomatis, Principal Investigator, MRC Human Nutrition Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HNR6480
Record Dates: First submitted 2017-08-07; First posted 2017-08-14 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Diet, Food, and Nutrition; Dietary Supplements
Keywords: polyphenols; green tea catechins; coffee caffeoylquinic acids; metabolism; inter-individual variability; colonic microbiota
MeSH Terms: interventions — Tea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Green tea and green coffee extract tablets — 1. Tablets: participants were required to take 6 green tea and 3 green coffee extract tablets daily for a period of 8 weeks. No tablets were taken during the last 4 weeks of the study. Randomly chosen tablets were analysed to quantify their polyphenol content.
  2. Urine collections: Several urine collections were required during the supplementation period in order have sufficient time points to estimate the plateau of the concentration of green tea and coffee polyphenols excreted in the urine to then be able to determine their bioavailability. There was a total of five 24-hour urine collections (at week 0 -before supplementation-, 2, 4, 8, and 12 -4 weeks after finishing the supplementation period).
  3. Completion of study documents: Participants were provided with urine collection sheets, polyphenol questionnaires, checklists to record polyphenol tablet intake, and detailed instructions.

SUMMARY:
There is little information on the dietary intake, absorption, metabolism and bioavailability (degree to which a substance becomes available to the target tissues upon administration) of polyphenols (natural substances present in a variety of foods) in human participants.

This study assessed the bioavailability in healthy participants of polyphenols from 2 supplements containing green tea and green coffee extracts.

Eleven participants were recruited and their habitual diet was assessed to estimate polyphenol intake. After completing a 24-hour urine collection, participants were given six green tea extract and three green coffee extract tablets, which they took daily for a period of 8 weeks. No tablets were taken during the last 4 weeks of the study. Further 24-hour urines were collected at 2, 4, 8 and 12 weeks.

Participants were required to attend HNR (medical laboratory) the day after each 24hour urine collection. At these visits, they were asked to bring along their urine collections, completed documents (urine collection sheet, checklist for tablet intake/side effects) and any remaining supplements, which were used to assess tablet compliance.

The investigators identified and quantified the amount of polyphenols in the supplement tablets as well as the amount of polyphenols and their metabolites in urine. The investigators then evaluated polyphenol bioavailability from the relationship between their dietary intake and urinary output.

Evidence from this research could inform future intervention studies by providing data on the bioavailability of green tea and coffee polyphenols, and on the individual differences related to phenolic intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women.
* 18-45 years of age.
* BMI between 18.5 and 24.9 kg/m2.

Exclusion Criteria:

* Smoking.
* Allergy or intolerance to intervention supplements.
* Chronic, acute or active inflammatory conditions, haematological disorders, or any other systemic illness of renal, hepatic or gastrointestinal origin.
* Major surgical operations in the gastrointestinal tract or medical treatment for gastrointestinal problems.
* Active cancer or diagnosis of malignancy within the last five years.
* Pregnant, lactating, contemplating pregnancy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2013-04-10 (Actual); Primary Completion 2013-10-18 (Actual); Study Completion 2013-10-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline phenolic metabolites in urine at 2 weeks | Week 0 -before supplementation- and week 2
  Assessment of the profile of metabolites coming from green tea and green coffee phytochemicals in urine
Change from baseline phenolic metabolites in urine at 4 weeks | Week 0 -before supplementation- and week 4
  Assessment of the profile of metabolites coming from green tea and green coffee
Change from baseline phenolic metabolites in urine at 8 weeks | Week 0 -before supplementation- and week 8
  Assessment of the profile of metabolites coming from green tea and green coffee
Change from baseline phenolic metabolites in urine at 12 weeks | Week 0 -before supplementation- and week 12 -4 weeks after finishing the supplementation period-
  Assessment of the profile of metabolites coming from green tea and green coffee

SECONDARY OUTCOMES:
Phenolic compounds in tablets | Through study completion, an average of 3 months
  Quantification of the tablet polyphenol content

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Tomatis, PhD, Principal Investigator — MRC HNR
Locations (1):
- MRC HNR Elsie Widdowson Laboratory, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No